CLINICAL TRIAL: NCT03340090
Title: Assessment of the Usefulness of Hemopatch in Coronary Artery Bypass Graft Surgery
Acronym: Hemopatch
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 022017
Record Dates: First submitted 2017-10-26; First posted 2017-11-13 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: CHD - Coronary Heart Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Two randomized groups of 100 patients will undergo standard CABG procedure in Cardio-Pulmonary Bypass (CPB). In first group (100 patients) two pieces of Hemopatch will be applied in one patient. Second group is the control group without above described intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (Experimental): First group of patients will undergo standard CABG procedure in CPB. In addition, two pieces of Hemopatch will be applied in one patient. One piece to improve hemostasis in the bed of left internal mammary artery (LIMA) harvesting and second piece of Hemopatch will be placed beneath the sternum.
  Interventions: Device: Medical Device Hemopatch-PEG-coated collagen patch
- Control (No Intervention): Second group of patients will undergo standard CABG procedure in CPB only.

INTERVENTIONS:
Device: Medical Device Hemopatch-PEG-coated collagen patch — Two pieces of PEG-coated collagen patch Hemopatch will be applied in one patient. One piece to improve hemostasis in the bed of LIMA harvesting and second piece of Hemopatch will be placed beneath the sternum.
  Arms: Intervention

SUMMARY:
The study aim is to assess polyethylene glycol (PEG) coated collagen patch (Hemopatch) on the quality of drainage after surgery, the length of hospital stay, the number of reoperations due to haemorrhage and treatment cost. The study will be conducted in 200 patients undergoing Coronary Artery Bypass Grafting (CABG) with the use of extracorporeal circulation and Internal mammary Artery (IMA) harvesting. Traditional method of haemostasis will be applied in 100 patients and Hemopatch will be additionally used in 100 subjects to prevent haemorrhage after IMA harvesting and sternum closure.

ELIGIBILITY:
Inclusion Criteria:

* coronary heart disease CHD (mammary harvesting)
* age>18
* informed consent

Exclusion Criteria:

* any condition that exclude patient from standard CABG procedure
* additional cardiac procedure to be conducted on subject in addition to CABG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Total postoperative drainage (ml) | measured 48 hours after surgery
  total amount of blood in the chest drainage system (mediastinum, pericardium, right and left pleura)
need for blood transfusion (number of blood units transfused) | measeured after surgery until hospital discharge (on avarage until 7th day after surgery)
  the total amount of blood passed to the patient
The number of reoperations | observed until 7 days after surgery
  The necessity of performing retoractomy due to excessive drainage or cardiac tamponade

SECONDARY OUTCOMES:
level of hemoglobin (g/dl) | after surgery until hospital discharge (on avarage until 7th day after surgery)
  level of hemoglobin tested in perioperative time frame
length of Intensive Care Unit stay (h) | on average 48 hours after surgery
  length of Intensive Care Unit stay measured in hours
hospital stay (days) | after surgery until hospital discharge (on average until 7th day after surgery)
  length of hospital stay after surgery
treatment cost (USD) | from patient hospital admission to hospital discharge ( on average 8-10 days)
  total treatment cost measured in both experimental and control group from hospital admission to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Michal Krejca, PhD, Md, Principal Investigator — Medical University of Lodz
Locations (1):
- Medical University of Lodz, Lodz, Łódź Voivodeship, Poland